CLINICAL TRIAL: NCT02991183
Title: A Feasibility Study of Acceptance and Commitment Therapy (ACT) to Promote the Wellbeing of Carers of People With Dementia
Brief Title: ACT for Carers of People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GN16MH672
Record Dates: First submitted 2016-12-02; First posted 2016-12-13 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2016-12

CONDITIONS: Dementia
Keywords: Caregivers; Acceptance and Commitment Therapy
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance and Commitment Therapy (Experimental): Two half day (2.5 hours) group ACT sessions delivered one week apart followed by a third session 2 weeks following the second session.
  Interventions: Behavioral: ACT

INTERVENTIONS:
Behavioral: ACT — A psychological therapy to help people i) notice and accept difficult thoughts and emotions; ii) identify what they value in life and iii) make changes to their behaviour to promote these values.

SUMMARY:
Background: Acceptance and Commitment Therapy (ACT) is a therapy that helps people to notice and accept difficult thoughts and emotions. ACT also helps people to identify what they value in life (e.g. a good relationship with their partner) and make changes to their behaviour to promote these values. Carers of people with dementia may experience reduced wellbeing associated with their role. Those whose wellbeing is greater than previously are said to be 'flourishing'.

Aim: The aim of this feasibility study is to evaluate the potential value of ACT as a group intervention for carers of people with dementia.

Methods: Participants will include adult carers of people with dementia. Study participants will be identified from two older people community mental health teams. Informed consent will be sought prior to group invitations being sent out. There will be two groups in total (12 in each group) and both groups will attend three 2.5 hour sessions of ACT. All participants will complete questionnaires at the beginning and 21 days later (asking questions about their thoughts and feelings, flourishing and about being a carer). Eight group participants will be invited to a focus group to understand what they found more helpful and less helpful.

Applications: Results from this study will potentially provide useful information to enable a further study with more participants to be conducted. The outcomes of this study will be shared with older people community mental health teams, dementia and carer specialist groups and potentially published in a relevant journal.

DETAILED DESCRIPTION:
Participants: two groups of participants will receive the ACT group intervention (Total n=24; n/Group = 12). One group of participants (n=8) who attend the ACT intervention will be invited to a focus group exploring intervention acceptability.

Recruitment Procedures: prior to recruitment commencing the researcher will present details of the study (recruitment procedures, eligibility criteria etc.) to the relevant Community Mental Health Teams (CMHTs) and at the Older Adult Psychology Team meeting. Carers of People with Dementia (CPwD) will be identified by National Health Service (NHS) staff working in Older People's CMHTs.

Potential participants will receive patient information sheet at routine appointments they attend with the person with dementia for whom they care. Carers will provide permission for their contact details to be passed to the research team using 'Notice of Interest' slip. The researcher will then arrange to meet with the carer to recruit them to the study. Informed consent will be sought and a member of the research team will complete a consent form with participants after they have had time to read the Participant Information Sheet. Consenting participants will be sent appointment letters with further details of the group.

Measures: participants will complete the following measures at the beginning and end of the ACT group intervention:

1. Demographic questionnaire (including age, gender, length of time being in a caring role, fulltime or part-time carers, any other employment, number of individuals they care for, and their relationship to the individual they care for (e.g. spouse, sibling, child, other).
2. Acceptance and Action Questionnaire: (AAQII). The AAQII is a 7 item questionnaire, which measures psychological flexibility on a 7 point Likert scale.
3. Mental Health Continuum-Short Form (MHC-SF). The MHC-SF is a 14 item questionnaire, measuring wellbeing on a 6 point Likert scale.
4. Experiential Avoidance in Caregiving Questionnaire (EACQ) The EACQ is a 15 item questionnaire, which measures experiential avoidance on a 5 point Likert scale.
5. Caregiver Burden Scale (CBS).The CBS is a 21 item questionnaire, which measures the overall level of burden carers experience in relation to their spouse or relative on a 5 point Likert scale.
6. Recruitment and retention parameters: A sample size of at least 12 people per group for pilot pharmaceutical studies will be an indicator of sufficient recruitment. However, 8 has been suggested as the optimum number of group participants in psychological interventions. Therefore, a figure of no more than 33% attrition from baseline to final assessment will be used to indicate that the ACT group intervention is feasible in terms of retention.
7. Group Evaluation Form: A brief survey will be completed with Likert scales and free text boxes for reflections on participants experience of attending the ACT groups.
8. Focus group: A smaller number of participants (n = 8) will also be invited to attend a focus group to explore their view of taking part in the ACT groups. This will be audio-recorded and transcribed for analysis.

Design: this project will be an uncontrolled feasibility trial, using convenience sampling, and measuring a range of variables pertinent to the feasibility of delivering ACT intervention groups for CPwD. Process evaluation methodology, including quantitative and qualitative methods, will be applied to measure feasibility of the group intervention and develop a greater understanding of the intervention delivered and its causal assumptions (see research questions above).

Quantitative data collected will include demographic information, number of participants recruited and retained throughout the study, outcome measures (carer burden, psychological flexibility, flourishing), and responses to Likert scale acceptability questions. Qualitative data will include responses to open-ended acceptability questions in the format of a questionnaire and focus group exploring participants' experience of attending the groups.

Research Procedures Measures will be completed by all participants at baseline (beginning of group) and 21 days post-baseline (end of group). Baseline measures will be completed prior to the first session. Post-baseline measures will be completed following the third session. Feedback surveys will be given to all participants at the last group session with Likert scales and free text boxes for reflections on their experience of attending the ACT groups.

A focus group of 8 participants who have completed the ACT group intervention will be conducted by a facilitator independent from the ACT group facilitators. The participants will be selected to provide a range of experiences of the group to elicit rich discussion and qualitative data regarding acceptability. A semi-structured interview will be used to guide discussions (including open questions related to group format and structure, ACT approach, practicalities of attending) but the participants will be encouraged to openly discuss their opinions of their experience of the ACT group.

ELIGIBILITY:
Inclusion Criteria:

* carers of people with a diagnosis of any type of dementia
* primary caregiver of the person with dementia for 3 months or more
* informed consent
* adequate English language skills

Exclusion Criteria:

* receiving any type of concurrent psychotherapy
* diagnosis of a severe or acute mental health problem (such as psychosis, anxiety, depression) when consent to participate is sought

Ages: 18 Years to 116 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited and retained to study completion | 4 weeks
Well-being | Time 0 and week 4
  Change in score from Mental Health Continuum Short Form questionnaire
Acceptability | 4 weeks
  Qualitative responses to Acceptability questionnaire devised by research team
Fidelity | 4 weeks
  Fidelity of the intervention to the ACT approach (measure developed by research team)

SECONDARY OUTCOMES:
Psychological Flexibility | Time 0 and week 4
  Change in score from Acceptance and Action Questionnaire-II
Psychological Flexibility in Caregivers | Time 0 and week 4
  Change in score from Experiential Avoidance in Caregiving Questionnaire
Caregiver Burden | Time 0 and week 4
  Change in score from Caregiver Burden Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hamish McLeod, PhD, Principal Investigator — University of Glasgow
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No